CLINICAL TRIAL: NCT01807078
Title: Randomized Comparison of the CHOlesterol-lowering Effects of nutraceuticaLs Versus Ezetimibe in Statin-intolerant patientS - The CHOLESS Trial
Brief Title: Cholesterol-lowering Effects of nutraceuticaLs Versus Ezetimibe in Statin-intolerant Patients
Acronym: CHOLESS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Pelliccia, Assistant Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 222-D-2013
Record Dates: First submitted 2013-03-06; First posted 2013-03-08 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ezetimibe; Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ezetimibe (Active Comparator): Patients will receive for 6 months ezetimibe (10 mg/day)
  Interventions: Drug: Ezetimibe
- Nutraceuticals (Active Comparator): Patients will receive for 6 months a commercially available nutraceutical combined pill (1 capsule/day containing monacolin K 10 mg, policosanol 10 mg, and phytosterols 300 mg
  Interventions: Dietary Supplement: Nutraceuticals

INTERVENTIONS:
Drug: Ezetimibe — 10 mg p.d. of ezetimibe
  Other Names: Zetia
  Arms: Ezetimibe
Dietary Supplement: Nutraceuticals — 1 capsule/day containing monacolin K 10 mg, policosanol 10 mg, and phytosterols 300 mg
  Other Names: Choless; Fixlipid
  Arms: Nutraceuticals

SUMMARY:
Treatment with statins has a class I indication after percutaneous coronary intervention (PCI), but is often discontinued by patients due to side effects.

Pharmacologic alternatives shown to be useful after PCI include ezetimibe and nutraceuticals (i.e. compounds derived from foods with cholesterol lowering actions).

It remains unknown, however, which of these two therapeutic approaches is more effective after PCI.

The primary objective of this study is to compare the efficacy and tolerability of ezetimibe vs. a nutraceutical-based protocol in statin-intolerant patients treated with percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background

Treatment with statins has a class I indication after percutaneous coronary intervention (PCI), but is often discontinued by patients due to side effects.

Pharmacologic alternatives shown to be useful after PCI include ezetimibe and nutraceuticals (i.e. compounds derived from foods with cholesterol lowering actions).

It remains unknown, however, which of these two therapeutic approaches is more effective after PCI.

Purpose

The primary objective of this study is to compare the efficacy and tolerability of ezetimibe vs. a nutraceutical-based protocol in statin-intolerant patients treated with percutaneous coronary intervention.

Study Population

Patients with coronary artery disease in stable conditions treated with percutaneous coronary intervention who have withdrawn statin treatment due to side effects

Randomization

Patients will be randomized to receive for 6 months either ezetimibe (10 mg/day) or a commercially available nutraceutical combined pill (1 capsule/day containing monacolin K 10 mg, policosanol 10 mg, and phytosterols 300 mg).

ELIGIBILITY:
Inclusion Criteria:

* Angiographically-proven coronary artery disease
* Recent (<12 months) percutaneous coronary intervention
* Class I indication to receive statin treatment
* Previous (<12 months) withdrawn of a statin due to side effects
* Unwilling to receive treatment with an alternative statin
* Able to understand and willing to sign the informed consent form

Exclusion Criteria:

• Women of child bearing potential patients must demonstrate a negative pregnancy test performed within 24 hours before CT

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reasons for treatment discontinuation | 6 months
  Reasons for treatment discontinuation

SECONDARY OUTCOMES:
Effects on lipid profile | 6 months
  Effects on cholesterol plasmatic levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University, Rome, Lazio, Italy